CLINICAL TRIAL: NCT01354080
Title: Comparison of the Effectiveness of Massage Based on the Tensegrity Rule and Classical Abdominal Massage in Persons With Constipation
Brief Title: The Effectiveness of Massage in Treating Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Marek Woźniewski, University School of Physical Education in Wroclaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03constip2011KASS
Record Dates: First submitted 2011-04-15; First posted 2011-05-16 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2010-03

CONDITIONS: Constipation
Keywords: constipation; massage; tensegrity
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- tensegrity massage (Experimental): In this group of patients massage sessions based on the tensegrity method were applied.
  Interventions: Other: massage based on the tensegrity rule
- classical massage (Active Comparator): In this group of patients classical massage sessions were applied
  Interventions: Other: massage - classical abdominal

INTERVENTIONS:
Other: massage based on the tensegrity rule — The massage consist of brushing the skin, stroking of the lower abdominal integuments. Elastic deformation of the thoracolumbar fascia. Then the abdominal integuments were elastically deformed by kneading to normalize the rest tension of the muscles of the abdominal integuments as well as, indirectly, the myofascial apparatus of the pelvic floor and in this way improve venous blood and lymph outflow from the large intestine and the sigmoid colon area. The next treatment stage - performing circular movements within the limits of the skin's mobility at 1/3 of the medial part of the thigh. By stroking movements in the direction of the armpit in accordance with the run of the thoracoepigastric and costalaxillary veins. Then the intercostal muscles were deformed.
  Arms: tensegrity massage
Other: massage - classical abdominal — The classical abdominal massage consisted of circular movements performed on the abdominal integuments by superficial and deep stroking techniques according to the colonic route (clockwise)
  Arms: classical massage

SUMMARY:
The purpose of this study is to compare the effectiveness of massage based on the tensegrity rule and classical abdominal massage in persons with constipation.

DETAILED DESCRIPTION:
Constipation can be defined as "an embarrassing ailment of the 21st century". It affects about 20-25% of the population, women as well as men, but occurs more frequently in women (female:male ratio of 2.2:1). Persons of different age suffer from it. Constipation is a bothersome ailment which negatively affects the general physical and mental state, lowers physical and mental fitness, significantly hinders professional work, and decreases life comfort As the factors which contribute to the occurrence of constipation are very diverse and complex, the treatment is a long-term and slow process. There are numerous conservative treatment methods for constipation, such as physical treatments, reflexotherapy, biofeedback, pharmacotherapy, and modification of lifestyle. There is also a possibility of applying classical massage in persons with constipation. However, observations of the authors suggest it is not a therapy commonly applied.

ELIGIBILITY:
Inclusion Criteria:

1. age from 18 to 70 years old
2. after therapy with Vermoks 2*1/ 3 regardless of body weight
3. negative Elis test for lambliasis
4. proper laboratory tests results: bilirubin, FA, GGTP, AspAT, AlAT
5. ultrasound scan of the abdominal cavity
6. positive interview based on questionnaire

Exclusion Criteria:

1. present cancer or prior cancer treatment, if there is no clear agreement of the involved oncologist
2. renal insufficiency > II NYHA
3. cardiovascular problems
4. respiratory insufficiency > II degree GOLD
5. unstable coronary disease
6. hypertensive crisis
7. liver insufficiency
8. prior liver transplant
9. prior or active hepatitis
10. jaundice
11. prior surgical treatments except: appendectomy >5 years before, cholecystectomy 5 years before
12. unequalized endocrinopathies
13. metabolic storage diseases
14. diabetes
15. nephrolithiasis
16. cholelithiasis
17. pancreatitis
18. chronic diseases of the intestines
19. diseases of the muscles
20. pregnancy
21. parasite infections of the digestive system (infection with human roundworm, lambliasis)
22. age above 18 years old
23. BMI> 33
24. improper ultrasound scan result or laboratory tests results
25. blood presence in feces

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-06; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Patient Questionnaire (including Rome Test) | baseline (immediately before the first massage session)
  The aims of the Patient Questionnaire were to proof constipation presence and supply evidence of the frequency and the quality of bowel movements, and to compare them with the state from Diary

SECONDARY OUTCOMES:
Diary of Bowel Movements | on 7th day and 21st day from the 1st massage session
  The aims of the Diary were to supply documentary evidence of the frequency and the quality of bowel movements, and to compare them with the state from before the experiment (the Patient Questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Kassolik, PhD, Study Chair — University School of Physical Education in Wrocław
Locations (1):
- University School of Physical Education in Wrocław, Wroclaw, Wroclaw Destrict, Poland

REFERENCES:
- [Background] Ingber DE. The architecture of life. Sci Am. 1998 Jan;278(1):48-57. doi: 10.1038/scientificamerican0198-48. PMID 11536845
- [Background] Kalish VB, Loven B, Sehgal M. Clinical inquiries. What is the best treatment for chronic constipation in the elderly? J Fam Pract. 2007 Dec;56(12):1050-2. No abstract available. PMID 18053448
- [Background] Kassolik K, Andrzejewski W, Trzęsicka E, Charlton G. Anatomical Grounds for the Use of the Tensegrity Principle in Massage. Fizjoterapia Polska 3(4) vol. 7: 332-343, 2007.
- [Background] Lamas K, Lindholm L, Stenlund H, Engstrom B, Jacobsson C. Effects of abdominal massage in management of constipation--a randomized controlled trial. Int J Nurs Stud. 2009 Jun;46(6):759-67. doi: 10.1016/j.ijnurstu.2009.01.007. Epub 2009 Feb 12. PMID 19217105
- [Background] Leung FW. Etiologic factors of chronic constipation: review of the scientific evidence. Dig Dis Sci. 2007 Feb;52(2):313-6. doi: 10.1007/s10620-006-9298-7. Epub 2007 Jan 12. PMID 17219073
- [Background] Stark ME. Challenging problems presenting as constipation. Am J Gastroenterol. 1999 Mar;94(3):567-74. doi: 10.1111/j.1572-0241.1999.00917.x. PMID 10086634
- [Background] Tariq SH. Constipation in long-term care. J Am Med Dir Assoc. 2007 May;8(4):209-18. doi: 10.1016/j.jamda.2007.02.009. PMID 17498603
- [Result] Ayas S, Leblebici B, Sozay S, Bayramoglu M, Niron EA. The effect of abdominal massage on bowel function in patients with spinal cord injury. Am J Phys Med Rehabil. 2006 Dec;85(12):951-5. doi: 10.1097/01.phm.0000247649.00219.c0. PMID 17117000
- [Result] Lacy BE. Defining and treating constipation in older adults. Am Fam Physician. 2006 Sep 1;74(5):715-6; author reply 716. No abstract available. PMID 16970017
- [Result] Bharucha AE. Constipation. Best Pract Res Clin Gastroenterol. 2007;21(4):709-31. doi: 10.1016/j.bpg.2007.07.001. PMID 17643910
- [Result] Chitkara DK, Talley NJ, Locke GR 3rd, Weaver AL, Katusic SK, De Schepper H, Rucker MJ. Medical presentation of constipation from childhood to early adulthood: a population-based cohort study. Clin Gastroenterol Hepatol. 2007 Sep;5(9):1059-64. doi: 10.1016/j.cgh.2007.04.028. Epub 2007 Jul 13. PMID 17632040
- [Result] Emly M. Abdominal massage. Nurs Times. 1993 Jan 20-26;89(3):34-6. No abstract available. PMID 8426818
- [Result] Harrington KL, Haskvitz EM. Managing a patient's constipation with physical therapy. Phys Ther. 2006 Nov;86(11):1511-9. doi: 10.2522/ptj.20050347. PMID 17079751
- [Result] Kassolik K, Andrzejewski W, Trzęsicka E. Role of the Tensegrity Rule in Theoretical Basis of Massage Therapy. Journal of Back and Musculoskeletal Rehabilitation 20(1):1053-8127, 2007.
- [Result] Kassolik K, Jaskolska A, Kisiel-Sajewicz K, Marusiak J, Kawczynski A, Jaskolski A. Tensegrity principle in massage demonstrated by electro- and mechanomyography. J Bodyw Mov Ther. 2009 Apr;13(2):164-70. doi: 10.1016/j.jbmt.2007.11.002. Epub 2007 Dec 21. PMID 19329052
- [Result] Klauser AG, Flaschentrager J, Gehrke A, Muller-Lissner SA. Abdominal wall massage: effect on colonic function in healthy volunteers and in patients with chronic constipation. Z Gastroenterol. 1992 Apr;30(4):247-51. PMID 1534955